CLINICAL TRIAL: NCT00046384
Title: Study of Aripiprazole in the Treatment of Patients With Acute Symptoms of Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Purpose: Treatment
Other Study IDs: CN138-077
Record Dates: First submitted 2002-09-27; First posted 2002-10-01 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2007-09

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — Aripiprazole

INTERVENTIONS:
Drug: aripiprazole

SUMMARY:
The purpose of this study is to learn if aripiprazole is effective in the treatment of patients with acute symptoms of Bipolar Disorder.

ELIGIBILITY:
Patients with acute symptoms of Bipolar Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-06; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (13):
  - Local Institution, Scottsdale, Arizona
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Chula Vista, California
  - Local Institution, Pico Rivera, California
  - Local Institution, Riverside, California
  - Local Institution, San Diego, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Winter Park, Florida
  - Local Institution, Staten Island, New York
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Nashville, Tennessee
  - Local Institution, Falls Church, Virginia
  - Local Institution, Bellevue, Washington
- Local Institution, Mendoza, Argentina